CLINICAL TRIAL: NCT00223288
Title: Caregiver Psychiatric Symptomatology and it's Relationship to Service Utilization by Children With Asthma
Brief Title: Impact of Caregiver Depression on Asthma in the Child
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sherwood Brown PI, UT Southwestern Medical Center at Dallas
Other Study IDs: MHGP MM12
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-08

CONDITIONS: Depressive Disorder, Major; Asthma
MeSH Terms: conditions — Depressive Disorder, Major; Asthma | interventions — Escitalopram

INTERVENTIONS:
Drug: Lexapro

SUMMARY:
This study will examine if depression in a primary caregiver is associated with more hospitalization or ER visits in children with asthma. This study will also explore whether treatment for depression in the primary caregivers is associated with improvement in asthma in school-aged children.

Asthma is a very common childhood disorder of airway inflammation. The causes include environmental irritants, cold temperature, and infection in the respiratory tract, and emotional factors can contribute to symptom exacerbation. However, asthma is a disease that can be well controlled if there is proper medication compliance and careful control of environmental conditions.

Data suggests that psychiatric symptoms in the mothers of children with asthma are associated with more asthma related hospitalizations in children. Thus, we want to explore this question further using more specific diagnostic instruments in order to detect what types of symptoms are associated with increased asthma related service utilization. Also, we want to explore if effective treatment of the caregivers' symptoms is associated with decreased hospitalization and emergency room visits for the child.

ELIGIBILITY:
Inclusion Criteria:

* Primary caregiver of a child currently hospitalized at Children's Medical Center of Dallas for an asthma exacerbation and between the ages of 5 and 16 years old
* Male and female
* English or Spanish Speaking
* Between the ages of 18 and 70 years old
* Caregivers with major depressive disorder will be offered treatment

Exclusion Criteria:

* At risk for suicide defined by multiple suicide attempts (greater than or equal to 3 in the past), and/or current suicidal ideation with a well-formed plan or intent
* Unlikely to attend follow-up appointments
* Mentally retarded or suffer from other severe cognitive impairment
* Pregnant or nursing, or women of childbearing age who will not use methods of birth control or abstinence during the study
* Suffering from a severe or life-threatening medical illness which would make completion of the study unlikely
* Suffering from treatment refractory depression defined by failing three adequate trials of antidepressants
* Depression as part of bipolar disorder or schizophrenia or schizoaffective disorder, or current depression secondary to a medication or general medical condition, or with psychotic features

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Primary caregiver of a child currently hospitalized at Children's Medical Center of Dallas for an asthma exacerbation and between the ages of 5 and 16 years old
Sampling Method: Non-Probability Sample
Enrollment: 175
Dates: Start 2003-03; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Sherwood Brown, MD, Ph.D., Principal Investigator — University of Texas, Southwestern Medical Center at Dallas
Locations (1):
- The University of Texas Southwestern Medical Center at Dallas, Dallas, Texas, United States